CLINICAL TRIAL: NCT01543217
Title: Use of a Respiratory Care Practitioner Disease Management (RCP-DM) Program for Patients Hospitalized With COPD
Brief Title: Respiratory Disease Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Barnes-Jewish Hospital (Other)
Responsible Party: Principal Investigator, Peggy Watts, Manager Respiratory Care Services, Barnes-Jewish Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 201201116
Record Dates: First submitted 2012-02-23; First posted 2012-03-02 (Estimated); Last update posted 2021-07-23 (Actual); Status verified 2016-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Active Comparator): Ususal care.
  Interventions: Other: Ususal care
- Intervention (Active Comparator): Patients assigned to the RT management arm will receive a 1-hour educational in-service conducted by a respiratory therapist case manager. The patient education session will include general information about COPD, direct observation of inhaler techniques, a review and adjustment of outpatient COPD medications, smoking cessation counseling, recommendations concerning influenza and pneumococcal vaccinations, encouragement of regular exercise, and instruction in hand hygiene.
  Interventions: Other: RT management

INTERVENTIONS:
Other: RT management — Patients assigned to the RT management arm will receive a 1-hour educational in-service conducted by a respiratory therapist case manager. The patient education session will include general information about COPD, direct observation of inhaler techniques, a review and adjustment of outpatient COPD medications, smoking cessation counseling, recommendations concerning influenza and pneumococcal vaccinations, encouragement of regular exercise, and instruction in hand hygiene.
  Arms: Intervention
Other: Ususal care — Routine respiratory care.
  Arms: Control

SUMMARY:
The aim of this study is to reduce the number of subsequent hospital admissions and/or emergency department (ED) visits for hospitalized patients with chronic obstructive pulmonary disease (COPD) by utilizing a respiratory care practitioner-led disease management (RCP-DM) program compared to standard discharge instructions and planning.

DETAILED DESCRIPTION:
The investigators propose to carry out a prospective, randomized, trial at Barnes-Jewish Hospital (1250-bed urban academic hospital). Eligible patients will be identified by a senior study coordinator who will also obtain informed consent for study participation. Adults greater than 18 years of age and less than 65 years of age will be eligible for enrollment if the lead investigator and the treating physician agree that the patient meets the enrollment criteria which include the following: patients with spirometrically confirmed COPD at high risk for repeat hospitalization or ED visits as predicted by hospital admission or ED visit in the previous 12 months for a COPD exacerbation, chronic home use of oxygen, or a course of systemic corticosteroid therapy in the preceding 12 months. Exclusion criteria include patients not expected to survive their hospitalization, presence of metastatic cancer, bed-bound individuals, non-English speaking patients, and patients unable to provide informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Adults greater than 18 years of age and less than 64 years of age will be eligible for enrollment if the lead investigator and the treating physician agree that the patient meets the enrollment criteria which include the following:

  * patients with spirometrically confirmed COPD at high risk for repeat hospitalization or emergency department (ED) visits as predicted by hospital admission or ED visit in the previous 12 months for a COPD exacerbation,
  * chronic home use of oxygen, or
  * a course of systemic corticosteroid therapy in the preceding 12 months.

Exclusion Criteria:

* patients not expected to survive their hospitalization,
* presence of metastatic cancer,
* bed-bound individuals,
* non-English speaking patients, and
* patients unable to provide informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 428 (Actual)
Dates: Start 2012-07; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The combined number of hospital admissions and ED visits for a COPD exacerbation | 6-month follow-up period
  Coordinators will use two strategies, First, they will monitor the automated medical record. All inpatient, outpatient, and ED visits to BJC affiliated institutions. Second coordinators will conduct bi-monthly telephone inquires to patients to determine if they had recent hospital or ED visits.

SECONDARY OUTCOMES:
Hospitalizations and ED visits for other causes | up to 3 months
  Number of times a subject is hospitalized or visit the ED during the study period.
Hospital and intensive care unit (ICU) lengths of stay | 6 months
  the number of days a subject is in the intensive care unit
Respiratory medication use | 6 months
  prescribed respiratory medications dose and usage
All causes of mortality | 6 months
  documentation of all causes of mortality

CONTACTS AND LOCATIONS:
Overall Officials: Marin Kollef, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Hospital, St Louis, Missouri, United States

REFERENCES:
- [Derived] Poot CC, Meijer E, Kruis AL, Smidt N, Chavannes NH, Honkoop PJ. Integrated disease management interventions for patients with chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2021 Sep 8;9(9):CD009437. doi: 10.1002/14651858.CD009437.pub3. PMID 34495549
- [Derived] Silver PC, Kollef MH, Clinkscale D, Watts P, Kidder R, Eads B, Bennett D, Lora C, Quartaro M. A Respiratory Therapist Disease Management Program for Subjects Hospitalized With COPD. Respir Care. 2017 Jan;62(1):1-9. doi: 10.4187/respcare.05030. Epub 2016 Nov 29. PMID 27899531